CLINICAL TRIAL: NCT03287882
Title: Prospective, Cluster Randomized Effectiveness Trial of Multiple Micronutrient Supplementation and Life Skills Education Provided From Preconception on Health and Nutrition Outcomes of Young, Reproductive-age Pakistani Women (15-24 Years)
Brief Title: Effect of Micronutrients and Life Skills Education on the Health and Nutrition of Adolescent and Young Women in Pakistan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); National Program for Family Planning and Primary Health Care (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Director, Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4324-Ped-ERC-16
Record Dates: First submitted 2017-08-21; First posted 2017-09-19 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Adolescents; Anemia; Pregnancy; Empowerment
Keywords: preconception supplementation; multiple micronutrients; low birth weight
MeSH Terms: conditions — Anemia; Empowerment | interventions — United Nations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Some investigators are blinded to the allocation of the intervention, and all study data collectors are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): 1. Preconception period: none
  2. Pregnancy period: daily iron (60 mg) and folic acid (400 µg) supplementation from confirmation of pregnancy; daily balanced energy protein supplements will additionally be provided to those participants who are underweight at the confirmation of pregnancy for the duration of the pregnancy
  3. Postpartum period: daily iron and folic acid supplementation to 6 months postpartum
- MMN supplementation and life skills education (Experimental): 1. Preconception period: twice-weekly MMN supplementation and bi-monthly group session including life skill based education materials
  2. Pregnancy period: daily MMN supplementation from confirmation of pregnancy; daily balanced energy protein supplements will additionally be provided to those participants who are underweight at the confirmation of pregnancy for the duration of the pregnancy
  3. Postpartum period: daily MMN supplementation to 6 months postpartum
  Interventions: Dietary Supplement: Multiple micronutrients (UNIMMAP composition); Behavioral: Life skills based education

INTERVENTIONS:
Dietary Supplement: Multiple micronutrients (UNIMMAP composition) — The intervention is an oral tablet containing 15 different vitamins and minerals at the UNIMMAP composition (includes 30 mg iron, 400 μg folic acid, 15 mg zinc, 2 mg copper, 65 μg selenium, 800 μg RE vitamin A, 1.4 mg vitamin B1, 1.4 mg vitamin B2, 18 mg niacin, 1.9 mg vitamin B6, 2.6 μg vitamin B12, 70 mg vitamin C, 5 μg vitamin D, 10 mg vitamin E and 150 μg iodine). Each tablet is small (approximately 10 mm diameter) and has been procured using the UNICEF supply catalogue. A single MMN supplementation dose will consist of a single tablet.
  Other Names: UNICEF, Micronutrient tabs, pregnancy/PAC-1000
  Arms: MMN supplementation and life skills education
Behavioral: Life skills based education — The life skills based education will be provided bi-monthly in the format of a group session throughout the preconception period. Three topic areas related to empowerment have been prioritized, including preventing early marriage; personal and menstrual hygiene practices; and the importance of nutrition to good health. Integrated within these topics will be messages related to the importance of continuing one's education, mental health, gender norms and equality, decision making, advocacy, resiliency, participation, communication skills, facing challenges, agency, conflict resolution, and the prevention of violence.
  Arms: MMN supplementation and life skills education

SUMMARY:
The primary aims of this study are: 1) To evaluate the impact of supplementation with multiple micronutrients (MMN) from preconception and life skills education among women 15-18.9 years of age at enrolment on the prevalence of anemia in a population setting; and 2) To evaluate the impact of supplementation with MMN from preconception and life skills education among young women 15-24 years of age on the rate of low birth weight (LBW) in a population setting. Infants born to mothers enrolled in the study will be followed for 1 year. This study aims to enrol 25,400 non-pregnant young women in Matiari district. This sample size is anticipated to equate to 1456 births. Participants will be randomized by cluster to receive either MMN supplements and life skills education or the standard of care at enrolment. Clusters have been defined based on health facility catchment areas. MMN supplements will be provided twice weekly during the preconception period, once daily during the pregnancy period, and once daily until 6 months after giving birth during the postpartum period; and a package of life skills education materials will be provided bi-monthly during the preconception period. In addition to the primary outcomes, measurements will include micronutrient status, anthropometrics, birth outcomes, dietary intake and feeding practices, adherence, and indices of empowerment.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age at enrolment: 15 years
* Maximum age at enrolment: 23 years
* Any marital status
* Intend to comply with study intervention and follow up

Exclusion Criteria:

* Women participating in other nutrition trials
* Women who intend to leave the study area
* Women who are already pregnant

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25447 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Anemia status | 0, 12*, 24 months (*in subgroup only)
  Hemoglobin concentration <12 g/dL
Low birth weight | At birth
  Birth weight <2500 g

SECONDARY OUTCOMES:
Biomarkers: serum ferritin, serum transferrin receptor, hepcidin, serum retinol, serum 25(OH)D, alpha-glycolytic protein, C-reactive protein (women) | Preconception (subgroup only): enrolment, 1 year, 2 years; Pregnancy: 4-12 weeks, 32 weeks; Postpartum: 1 week
Anthropometrics: height (women) | Preconception: enrolment, 6 months*, 1 year, 2 years (*in subgroup only); Pregnancy: 4-12 weeks, 32 weeks; Postpartum: 1 week, 6 months
Anthropometrics: middle upper arm circumference (women) | Preconception: enrolment, 6 months*, 1 year, 2 years (*in subgroup only); Pregnancy: 4-12 weeks, 32 weeks; Postpartum: 1 week, 6 months
Anthropometrics: weight (women) | Preconception: enrolment, 6 months*, 1 year, 2 years (*in subgroup only); Pregnancy: 4-12 weeks, 32 weeks; Postpartum: 1 week, 6 months
Gestational age | At birth
Preterm birth | At birth
Stillbirth | At birth
Small for gestational age | At birth
Birth size: length | Within 24 hours of birth
Birth size: head circumference | Within 24 hours of birth
Birth size: middle upper arm circumference | Within 24 hours of birth
Birth size: weight | Within 24 hours of birth
Birth defects | At birth
Infant growth: length | 1, 3, 6, 9, 12 months
Infant growth: head circumference | 1, 3, 6, 9, 12 months
Infant growth: middle upper arm circumference | 1, 3, 6, 9, 12 months
Infant growth: weight | 1, 3, 6, 9, 12 months
Age at marriage | Enrolment, 1 year, 2 years
Completion of 10th grade education | Enrolment, 1 year, 2 years
Use of sanitary pad during last menstrual period | Enrolment, 1 year, 2 years
Dietary intake: 24-hour recall (subgroup of women) | Preconception: enrolment; Pregnancy: 4-12 weeks, 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar A Bhutta, PhD, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Matiari Research and Training Centre, Matiari, Sindh, Pakistan

REFERENCES:
- [Derived] Baxter JB, Wasan Y, Daniel AI, Begum K, Hussain A, Iqbal J, Aufreiter S, Beggs MR, Duan L, Greco A, Huang C, Soofi S, Bandsma RH, Bhutta ZA, O'Connor DL. Maternal multiple micronutrient supplementation in rural Pakistan increased some milk micronutrient concentrations, but not infant growth, at three-months postpartum: a randomized controlled trial substudy. Am J Clin Nutr. 2025 Jul;122(1):174-184. doi: 10.1016/j.ajcnut.2025.05.019. Epub 2025 May 21. PMID 40409469
- [Derived] Baxter JB, Wasan Y, Hussain A, Soofi SB, Ahmed I, Bhutta ZA. Drivers of malnutrition among late adolescent and young women in rural Pakistan: a cross-sectional assessment of the MaPPS trial. BMJ Open. 2023 May 23;13(5):e063734. doi: 10.1136/bmjopen-2022-063734. PMID 37221027
- [Derived] Baxter JB, Kortenaar JL, Wasan Y, Hussain A, Soofi SB, Ahmed I, Bhutta ZA. Age-Based Anthropometric Cutoffs Provide Inconsistent Estimates of Undernutrition: Findings from a Cross-Sectional Assessment of Late-Adolescent and Young Women in Rural Pakistan. Curr Dev Nutr. 2021 Nov 10;5(11):nzab130. doi: 10.1093/cdn/nzab130. eCollection 2021 Nov. PMID 34901693
- [Derived] Bhutta ZA. Reply to NF Krebs and KM Hambidge. Am J Clin Nutr. 2019 Aug 1;110(2):521-522. doi: 10.1093/ajcn/nqz078. No abstract available. PMID 31367763
- [Derived] Bhutta ZA. Balancing the benefits of maternal nutritional interventions; time to put women first! Am J Clin Nutr. 2019 Feb 1;109(2):249-250. doi: 10.1093/ajcn/nqy336. No abstract available. PMID 30721972
- [Derived] Baxter JB, Wasan Y, Soofi SB, Suhag Z, Bhutta ZA. Effect of life skills building education and micronutrient supplements provided from preconception versus the standard of care on low birth weight births among adolescent and young Pakistani women (15-24 years): a prospective, population-based cluster-randomized trial. Reprod Health. 2018 May 31;15(1):104. doi: 10.1186/s12978-018-0545-0. PMID 29855317
- [Derived] Baxter JB, Wasan Y, Soofi SB, Suhag Z, Bhutta ZA. Feasibility and effect of life skills building education and multiple micronutrient supplements versus the standard of care on anemia among non-pregnant adolescent and young Pakistani women (15-24 years): a prospective, population-based cluster-randomized trial. Reprod Health. 2018 May 30;15(1):103. doi: 10.1186/s12978-018-0547-y. PMID 29848335